CLINICAL TRIAL: NCT04495309
Title: Effectiveness and Tolerability of Metastases-directed Radiotherapy in Addition to Standard Systemic Therapy in Patients With Oligometastatic Breast Cancer: A Randomized Controlled Multinational and Multicenter Clinical Trial
Brief Title: Metastases-directed Radiotherapy in Addition to Standard Systemic Therapy in Patients With Oligometastatic Breast Cancer
Acronym: OLIGOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARO-2015-1
Record Dates: First submitted 2020-06-09; First posted 2020-07-31 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Oligometastatic Breast Cancer; Radiotherapy; Progression-free survival (PFS)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Standard of care, i. e. no local radiotherapy in addition to standard systemic therapy (exception: palliative local treatment of symptomatic lesions where indicated)
- Experimental (Experimental): Standard of care (standard systemic therapy) + study intervention
  Interventions: Radiation: Metastases-directed Radiotherapy

INTERVENTIONS:
Radiation: Metastases-directed Radiotherapy — Ablative radiotherapy (radiosurgery, stereotactic radiotherapy, hypofractionated image-guided radiotherapy (IGRT)) with few high-dose fractions
  Arms: Experimental

SUMMARY:
The prognosis for patients with metastatic breast cancer has improved continuously. Systemic therapies alone are not able to cure the disease permanently.

Investigators initiated this randomized controlled multinational and multicenter clinical trial to analyse the impact of a local metastases-directed radiotherapy in addition to standard systemic therapy in patients with oligometastatic breast cancer on progression-free survival and quality of life.

DETAILED DESCRIPTION:
Preferably ablative radiotherapy (radiosurgery, stereotactic radiotherapy, hypofractionated image-guided radiotherapy (IGRT)) with few high-dose fractions. Larger lesions or lesions with critical normal tissue involvement should be treated with three-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) in moderate hypofractionated radiotherapy (depending on the size and location of the target volume and the decision of the radiooncologist). For critical organs in the target volume, standard fractionated radiotherapy can be used.

ELIGIBILITY:
Inclusion Criteria:

* Metastasized breast cancer - up to 5 clinically manifest (new, progressive, persistent) metastases (a lymph node metastasis and a circumscribed local recurrence are each considered as one metastasis, i.e. also locoregional recurrent breast carcinomas with additional hematogenic metastasis possible)
* maximum of 3 cerebral metastases known
* indication for palliative drug therapy (endocrine therapy and/or chemotherapy and/or treatment with other substances) given according to guidelines (1st-line or further therapy lines, a special regime is not specified)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* local radiation of all metastases possible
* presentation of a written declaration of consent
* patient ≥ 18 years

Exclusion Criteria:

* Previous radiotherapy, if this interferes with treatment within the scope of the study
* symptomatic metastases requiring local therapy of all metastases (e.g. pain radiation), a radiation indication (or other local therapy) for individual metastases is not a criterion for exclusion
* known central nervous system (CNS) metastasis without extracerebral metastasis (in these cases, immediate local therapy is mandatory)
* more than three known CNS metastases (no indication for purely local therapy of only the metastases, primary whole brain radiation is indicated)
* multifocal metastasis in one organ with impossibility to comply with the dose constraints for this organ (e.g., no indication for local therapy of only the metastases, primary whole brain radiation is indicated) (e.g. in the liver)
* exclusively regional lymph node metastasis without haematogenic metastases (in these cases local therapy is clearly indicated according to guidelines)
* relevant comorbidity, if this results in restrictions for further therapy
* Incapacity to contract or lack of informed consent
* Pregnancy and lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with oligometastatic breast cancer
Enrollment: 564 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
First co-primary outcome measure is progression-free survival (PFS) | at least 12 months after randomization
  Co-primary progression-free survival (PFS) according to Response Evaluation Criteria In Solid Tumors (RECIST)
Second co-primary outcome measure is quality of life | 12 weeks after randomization
  Co-primary quality of life according to European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Cancer patients with 30 items (QLQ-C30) sum score

SECONDARY OUTCOMES:
Feasibility (per-protocol within intention-to-treat) | 12 weeks
  Proportion of participants treated per protocol
Overall survival | at least 1, up to 5 years
  Time between randomization and death
Toxicity (number and degree of reported toxicities in both treatment arms) | 0 to 5 years
  Proportion of participants with degree of toxicities as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) and by Radiation Treatment Oncology Group (RTOG) by point in time of follow-up with higher degree indicating higher intensity
Neoplasia-specific quality of life | quarterly up to 5 years
  Research and Treatment of Cancer (EORTC) Quality of Life Questionaire for Cancer patients with 30 items (QLQ-C30) with different scales
Breast cancer-specific quality of life | quarterly up to 5 years
  Research and Treatment of Cancer (EORTC) Quality of Life Questionaire for breast cancer patients with 23 items (QLQ-BR23) on 4-point Likert scales with different directions
Patient satisfaction | 12 weeks
  Research and Treatment of Cancer (EORTC) Patient satisfaction questionnaire for cancer patients with 33 items (PATSAT-C33) on 5-point Likert scale with higher scores indicating greater satisfaction
Frequency of adverse events | 0 to 5 years
  Number of patients with adverse and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Dunst, Professor, Study Director — University Hospital Schleswig-Holstein
Locations (14):
- Germany (14):
  - Universitätsmedizin Mannheim Klinik für Strahlentherapie und Radioonkologie, Mannheim, Baden-Wurttemberg
  - Praxis für Strahlentherapie und Radioonkologie am Krankenhaus Weilheim, Weilheim, Bavaria
  - Klinikum Frankfurt (Oder) GmbH Klinik für Strahlentherapie/Radioonkologie, Frankfurt (Oder), Brandenburg
  - Universitätsklinikum Marburg Klinik für Strahlentherapie und Radioonkologie, Marburg, Hesse
  - GSR Hameln im Sana Klinikum Hameln-Pyrmont, Hamelin, Lower Saxony
  - Gemeinschaftspraxis für Strahlentherapie, Hildesheim, Lower Saxony
  - MVZ WOB GmbH Strahlentherapie, Wolfsburg, Lower Saxony
  - Strahlentherapie Bocholt Gemeinschaftspraxis und Belegabteilung am St.-Agnes-Hospital, Bocholt, North Rhine-Westphalia
  - Evangelische Kliniken Gelsenkirchen Klinik für Strahlentherapie, Gelsenkirchen, North Rhine-Westphalia
  - Xcare Praxis für Strahlentherapie Saarlouis am Marienkrankenhaus, Saarlouis, Saarland
  - Städtisches Klinikum Dresden, Strahlentherapie, Dresden, Saxony
  - Heinrich-Braun-Klinikum Zwickau gGmbH Klinik für Strahlentherapie und Radioonkologie, Zwickau, Saxony
  - Christian-Albrechts-University Kiel, University Medical Center Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal

REFERENCES:
- [Derived] Krug D, Vonthein R, Illen A, Olbrich D, Barkhausen J, Richter J, Klapper W, Schmalz C, Rody A, Maass N, Bauerschlag D, Hessler N, Konig IR, Dellas K, Dunst J. Metastases-directed Radiotherapy in Addition to Standard Systemic Therapy in Patients with Oligometastatic Breast Cancer: Study protocol for a randomized controlled multi-national and multi-center clinical trial (OLIGOMA). Clin Transl Radiat Oncol. 2021 Apr 5;28:90-96. doi: 10.1016/j.ctro.2021.03.012. eCollection 2021 May. PMID 33912695